CLINICAL TRIAL: NCT03728972
Title: Pilot Study of Pembrolizumab in Untreated Extranodal, NK/T Cell Lymphoma, Nasal Type
Brief Title: Study of Pembrolizumab in Patients With Early-Stage NK/T-cell Lymphoma, Nasal Type
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-393
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: NK/T-Cell Lymphoma of Nasal Cavity (Diagnosis); NK/T-Cell Lymphoma of Nasopharynx (Diagnosis)
Keywords: Pembrolizumab; Early stage NK/T-Cell Lymphoma; 18-393; Memorial Sloan kettering Cancer Center
MeSH Terms: conditions — Disease | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) (Experimental)
  Interventions: Drug: Pembrolizumab
- Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV) (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IVPB every 3 weeks

SUMMARY:
The purpose of this study is to test how well pembrolizumab shrinks Early-Stage NK/T-cell Lymphoma (ENKTL) in participants who have not yet received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of extranodal NK/T, nasal type cell lymphoma at the enrolling institution
* 18 years of age on day of signing informed consent
* Have a performance status of ≤ 1 on the ECOG Performance Scale
* Have measurable disease by PET/CT
* Demonstrate adequate organ function as defined below:

RENAL:

Serum Creatinine ≤ 1.5 x upper limit of normal (ULN)

OR

Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCL) Serum creatinine ≥ 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN ≤ 1.5 x upper limit of normal (ULN)

OR

Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCL) ≥ 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN

HEPATIC:

Serum total bilirubin ≤ 1.5 x ULN

OR

Serum total bilirubin ≤ 3 x ULN for subjects with liver metastases

AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN

OR

AST (SGOT) and ALT (SGPT) ≤ 5 x ULN for subjects with liver metastases

CARDIAC:

Ejection fraction ≥ 50%

PULMONARY:

Hemoglobin-adjusted diffusing capacity for carbon monoxide ≥ 50%

- Women of childbearing potential* must have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to receiving the first dose of study medication

* *A woman of childbearing potential is a sexually mature female who has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months)

  * Women of childbearing potential must be willing to use an adequate method of contraception
* Must agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 120 days after the last dose of study therapy, or agree to completely abstain from heterosexual intercourse

  * Male subjects of childbearing potential must agree to use an adequate method of contraception
* Male subjects, even if surgically sterilized (i.e. statue post vasectomy) must agree to 1 of the following: Practice effective barrier contraception during the entire study therapy, or agree to completely abstain from heterosexual intercourse

Exclusion Criteria:

* Received prior treatment for extranodal NK/T cell lymphoma
* Medical illness unrelated to lymphoma, which, in the opinion of the treating physician and/or institutional principal investigator, makes participation in this study inappropriate.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has active Hepatitis B (defined as HBV DNA is detected) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2026-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Stanford University, Stanford, California
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Md Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV)
Started | 15 | 4
Completed | 6 | 1
Not Completed | 9 | 3
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Disease progression | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV) | Total
Number analyzed (Participants) | 15 | 4 | 19
Age, Continuous [Median (Full Range); unit: years] | 53 [40 to 83] | 43.5 [19 to 64] | 53 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 10 | 2 | 12
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 2 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate of Pembrolizumab in Untreated Early-Stage NK/T-cell Lymphoma, Nasal Type (ENKTL)
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of pts with complete response
Arm/Group | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV)
Number analyzed (Participants) | 15 | 4
percentage of pts with complete response | 47 [21 to 73] | 25 [1 to 81]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV)
All-Cause Mortality (participants affected / at risk) | 4/15 | 2/4
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/4
Other Adverse Events (participants affected / at risk) | 14/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) (N=15) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV) (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage I/II) (N=15) | Early-Stage NK/T-cell Lymphoma/ENKTL (Stage III/IV) (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epigastric Pain (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 6 | 2
Fever (General disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Herpetic Lesion - Lip (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Itchy Lip Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Itchy Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Lipase increased (Investigations) | 2 | 0
Localized edema (General disorders) | 1 | 0
Mild Cold (General disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Nose Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
papulopustular rash extremities and torso (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Serum amylase increased (Investigations) | 2 | 0
Skin Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sores on Upper Palate (Gastrointestinal disorders) | 1 | 0
Thyroid Stimulating Hormone Increased (Investigations) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary pressure (Renal and urinary disorders) | 1 | 0
LFTs elevated (Hepatobiliary disorders) | 6 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
erythematous red spot on shoulder, scalp, and torso (Skin and subcutaneous tissue disorders) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Mild erythematous rash on torso (Skin and subcutaneous tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03728972/Prot_SAP_000.pdf